CLINICAL TRIAL: NCT00049829
Title: HORIZON-PFT: Pivotal Fracture Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CZOL446H2301
Record Dates: First submitted 2002-11-14; First posted 2002-11-15 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-11

CONDITIONS: Osteoporosis
Keywords: Bisphosphonate,BMD,Height loss, Hip protectors,HRT,; Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Zoledronic Acid

INTERVENTIONS:
Drug: Zoledronic Acid

SUMMARY:
HORIZON-PFT (Pivotal Fracture Trial) will study the effect of zoledronic acid, given once per year, on the treatment of osteoporosis in women past menopause. Hip and vertebral fractures are the most devastating consequences of osteoporosis. HORIZON-PFT is designed to determine the benefits of zoledronic acid in fracture reduction at both the hip and spine.

ELIGIBILITY:
Inclusion Criteria:

* Female, 65-89 years old
* No history of severe liver, kidney or eye disease

Exclusion Criteria:

* Current bisphosphonate users such as Aredia® (pamidronate), Didronel® (etidronate), Fosamax® (alendronate), Actonel® (risedronate), Skelid® (tiludronate)
* Using hip protectors

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 65 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 7700
Dates: Start 2002-01; Primary Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Incidence of hip fxs
Incidence of new vertebral fxs

SECONDARY OUTCOMES:
Percent change in hip BMD
New and/or worsening vertebral fxs
All clinical fxs

CONTACTS AND LOCATIONS:
Locations (60):
- United States (59):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Arthritis Research, Paradise Valley, Arizona
  - Southern Arizona VA, Tucson, Arizona
  - University of Arkansas for Medical Science, Little Rock, Arkansas
  - Osteoporosis Medical Center, Beverly Hills, California
  - Orthopaedic Hospital, Los Angeles, California
  - The Foundation for Osteoporosis Research and Education, Oakland, California
  - University of California Davis- Gen Med Research, Sacramento, California
  - Osteoporosis Prevention Center, San Diego, California
  - Radiant Research- San Diego, San Diego, California
  - Diablo Clinical Research, Inc, Walnut Creek, California
  - Colorado Center for Bone Research, Lakewood, Colorado
  - Longmont Medical Research Network, Longmont, Colorado
  - Northeast Clinical Research, Hamden, Connecticut
  - Health Core, Newark, Delaware
  - CRA Research, Fort Lauderdale, Florida
  - Anchor Research Center, Naples, Florida
  - Sarasota Arthritis Center, Sarasota, Florida
  - Radiant, Stuart, Florida
  - Comprehensive Clinical Trials, LLC, West Palm Beach, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - United Osteoporosis Centers (UOC), Gainesville, Georgia
  - Northwestern University Center for Clinical Research, Chicago, Illinois
  - School of Medicine, Indianapolis, Indiana
  - Medical Specialists, Munster, Indiana
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Center for Arthritis and Osteoporosis, Elizabethtown, Kentucky
  - Maine Center for Osteoporosis Research and Education, Bangor, Maine
  - Osteoporosis Clinical Trial Center, Hagerstown, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Clinical Pharmacology Study Groups, Worcester, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Arthritis Regional Research Center, Mercerville, New Jersey
  - Phoenix OB-GYN Associates, LLC, Moorestown, New Jersey
  - New Mexico Clinical Research and Osteoporosis Center, Inc, Albuquerque, New Mexico
  - Endwell Family Physicians, Endwell, New York
  - Winthrop U Hospital, Mineola, New York
  - Internal Medicine Associates, Fargo, North Dakota
  - University of Cincinnati Bone Health and Osteoporosis Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Einstein, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Radiant, Wyomissing, Pennsylvania
  - Rhode Island Hospital, Osteoporosis Research/ Bone Density Unit, Providence, Rhode Island
  - Roger William Medical Center, Providence, Rhode Island
  - Avera Research Institute, Sioux Falls, South Dakota
  - University of Tennessee Health Science, Memphis, Tennessee
  - West Cancer Clinic, Memphis, Tennessee
  - Diabetes Regional Research Center, Midland, Texas
  - Sam Clinical Research Center, San Antonio, Texas
  - University of Texas Health Center at Tyler -Center for Clinical Research, Tyler, Texas
  - Hampton Roads Center for Clinical Research, Inc, Norfolk, Virginia
  - McGuire Veterans Affairs Medical Center, Richmond, Virginia
  - VA Commonwealth University, Richmond, Virginia
  - Osteoporosis Research Unit, Seattle, Washington
  - The Physicians Clinic, Spokane, Washington
- Novartis, Nuremberg, Germany

REFERENCES:
- [Derived] Cai G, Keen HI, Host LV, Aitken D, Laslett LL, Winzenberg T, Wluka AE, Black D, Jones G. Once-yearly zoledronic acid and change in abdominal aortic calcification over 3 years in postmenopausal women with osteoporosis: results from the HORIZON Pivotal Fracture Trial. Osteoporos Int. 2020 Sep;31(9):1741-1747. doi: 10.1007/s00198-020-05430-z. Epub 2020 May 2. PMID 32361951
- [Derived] Mathew A, Brufsky A. Bisphosphonates do not reduce breast cancer in postmenopausal women. Ann Intern Med. 2015 Jan 20;162(2):JC5. doi: 10.7326/ACPJC-2015-162-2-005. No abstract available. PMID 25599365
- [Derived] Hue TF, Cummings SR, Cauley JA, Bauer DC, Ensrud KE, Barrett-Connor E, Black DM. Effect of bisphosphonate use on risk of postmenopausal breast cancer: results from the randomized clinical trials of alendronate and zoledronic acid. JAMA Intern Med. 2014 Oct;174(10):1550-7. doi: 10.1001/jamainternmed.2014.3634. PMID 25111880
- [Derived] Cauley JA, Black D, Boonen S, Cummings SR, Mesenbrink P, Palermo L, Man Z, Hadji P, Reid IR; HORIZON Pivotal Fracture Group. Once-yearly zoledronic acid and days of disability, bed rest, and back pain: randomized, controlled HORIZON Pivotal Fracture Trial. J Bone Miner Res. 2011 May;26(5):984-92. doi: 10.1002/jbmr.292. PMID 21542001
- [Derived] Grbic JT, Black DM, Lyles KW, Reid DM, Orwoll E, McClung M, Bucci-Rechtweg C, Su G. The incidence of osteonecrosis of the jaw in patients receiving 5 milligrams of zoledronic acid: data from the health outcomes and reduced incidence with zoledronic acid once yearly clinical trials program. J Am Dent Assoc. 2010 Nov;141(11):1365-70. doi: 10.14219/jada.archive.2010.0082. PMID 21037195
- [Derived] Eastell R, Black DM, Boonen S, Adami S, Felsenberg D, Lippuner K, Cummings SR, Delmas PD, Palermo L, Mesenbrink P, Cauley JA; HORIZON Pivotal Fracture Trial. Effect of once-yearly zoledronic acid five milligrams on fracture risk and change in femoral neck bone mineral density. J Clin Endocrinol Metab. 2009 Sep;94(9):3215-25. doi: 10.1210/jc.2008-2765. Epub 2009 Jun 30. PMID 19567517
- [Derived] Black DM, Delmas PD, Eastell R, Reid IR, Boonen S, Cauley JA, Cosman F, Lakatos P, Leung PC, Man Z, Mautalen C, Mesenbrink P, Hu H, Caminis J, Tong K, Rosario-Jansen T, Krasnow J, Hue TF, Sellmeyer D, Eriksen EF, Cummings SR; HORIZON Pivotal Fracture Trial. Once-yearly zoledronic acid for treatment of postmenopausal osteoporosis. N Engl J Med. 2007 May 3;356(18):1809-22. doi: 10.1056/NEJMoa067312. PMID 17476007